CLINICAL TRIAL: NCT01911182
Title: A Prospective, Controlled Trial of Inhalation of Low Concentration of CO2 in Preterm Infants Not Responding to Caffeine for the Treatment of Apnea of Prematurity
Brief Title: Inhalation of Low Concentration of CO2 in Preterm Infants Not Responding to Caffeine for the Treatment of Apnea
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Institute of Child Health (Industry)
Responsible Party: Principal Investigator, Ruben Alvaro, Associate Professor of Pediatrics, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B2011:072
Record Dates: First submitted 2011-09-22; First posted 2013-07-30 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Apnea of Prematurity
Keywords: apnea of prematurity; control of breathing; newborn; CO2 inhalation
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhalation of low concentration of CO2 (Experimental)
  Interventions: Other: Inhalation of low concentration of CO2
- caffeine only (Active Comparator)
  Interventions: Other: Inhalation of low concentration of CO2

INTERVENTIONS:
Other: Inhalation of low concentration of CO2 — Inhalation of 1% CO2 through nasal prongs
  Other Names: Inhalatio of biological gas

SUMMARY:
In premature infants, apnea of prematurity is one of their major clinical problems. Caffeine is currently a worldwide therapy to reduce the number and severity of these apneas. This practice has shown to be safe on cognitive and neurodevelopmental outcomes at 18 to 21 months of age. However, caffeine is not 100% effective, and may have little effect on hypoxemia and bradycardia. Infants with intractable apneas unresponsive to caffeine treatment may require endotracheal intubation and mechanical ventilation. This procedure is invasive and has been associated with complications and increased risk for chronic lung disease and adverse neurodevelopmental outcome. Therefore, an alternative treatment modality would be preferable if it would prevent the infants from requiring endotracheal intubation. The investigators have been testing the overall hypothesis that small concentrations of inhaled CO2 (~1%) are effective in treating apnea of prematurity. The investigators have completed three studies in preterm infants showing that inhalation of low concentration of CO2, in infants not on caffeine, regularize breathing and decrease apneas significantly. The effects of inhalation of CO2 in infants already on caffeine, are unknown. The hypothesis to be tested is that inhalation of low concentration CO2 (1%) will significantly reduce apnea in infants treated with caffeine. The investigators have three specific aims in this proposal. 1) the investigators want to know if the apnea rate (number of apneas of ≥5 seconds/hour) is decreased with CO2 inhalation in preterm infants already on caffeine for the treatment of apnea of prematurity; 2) the investigators want to know whether inhalation of CO2 can make breathing more regular with less apneic time and whether it decreases prolonged apneas (>20 seconds) in infants already on caffeine for the treatment of apnea of prematurity; 3) the investigators want to assess the effect of inhalation of low concentration of CO2 on the regional oxygen saturation of the brain measured by near-infrared spectroscopy (NIRS) during apneas. This is to see whether CO2, by protecting cerebral blood flow, minimizes the decrease in cerebral oxygenation during apneas. This study entails a new and possibly more physiological method of treating apneas of prematurity that can be added to the present treatment of caffeine. These two treatments together, could minimize the number and severity of apneas and possibly decrease the need for mechanical ventilation in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth < 33 weeks
* on caffeine treatment for apnea of prematurity at a maintenance dose of 5 mg/kg/day
* having apnea of prematurity (at least 5 self-resolved apneas or 2 apneas requiring intervention/12 hours)

Exclusion Criteria:

* on mechanical ventilation
* presence of congenital anomalies, sepsis or other known causes of apnea
* failure to obtain parental consent

Ages: 3 Days to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Effect of inhalation of low concentration of CO2 (1%) on the apnea rate (number of apneas of ≥5 seconds/hour) in preterm infants already on caffeine for the treatment of apnea of prematurity. | 3 hours

SECONDARY OUTCOMES:
Effect of low concentration of CO2 on apneic time in seconds per hour and duration of long apneas in seconds | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ruben E Alvaro, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Al-Saif S, Alvaro R, Manfreda J, Kwiatkowski K, Cates D, Qurashi M, Rigatto H. A randomized controlled trial of theophylline versus CO2 inhalation for treating apnea of prematurity. J Pediatr. 2008 Oct;153(4):513-8. doi: 10.1016/j.jpeds.2008.04.025. Epub 2008 Jun 4. PMID 18534618
- [Background] Al-Aif S, Alvaro R, Manfreda J, Kwiatkowski K, Cates D, Rigatto H. Inhalation of low (0.5%-1.5%) CO2 as a potential treatment for apnea of prematurity. Semin Perinatol. 2001 Apr;25(2):100-6. doi: 10.1053/sper.2001.23199. PMID 11339662
- [Background] Alvaro RE, Khalil M, Qurashi M, Al-Saif S, Al-Matary A, Chiu A, Minski J, Manfreda J, Kwiatkowski K, Cates D, Rigatto H. CO(2) inhalation as a treatment for apnea of prematurity: a randomized double-blind controlled trial. J Pediatr. 2012 Feb;160(2):252-257.e1. doi: 10.1016/j.jpeds.2011.07.049. Epub 2011 Sep 9. PMID 21907349
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW; Steering Committee of the Caffeine for Apnea of Prematurity (CAP) trial. Archimedes: Does caffeine treatment for apnoea of prematurity improve neurodevelopmental outcome in later life? Arch Dis Child. 2011 Aug;96(8):784. doi: 10.1136/adc.2010.206698. Epub 2011 Mar 4. No abstract available. PMID 21377992
- [Background] Davis PG, Schmidt B, Roberts RS, Doyle LW, Asztalos E, Haslam R, Sinha S, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine for Apnea of Prematurity trial: benefits may vary in subgroups. J Pediatr. 2010 Mar;156(3):382-7. doi: 10.1016/j.jpeds.2009.09.069. Epub 2009 Nov 18. PMID 19926098
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Long-term effects of caffeine therapy for apnea of prematurity. N Engl J Med. 2007 Nov 8;357(19):1893-902. doi: 10.1056/NEJMoa073679. PMID 17989382
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine therapy for apnea of prematurity. N Engl J Med. 2006 May 18;354(20):2112-21. doi: 10.1056/NEJMoa054065. PMID 16707748